CLINICAL TRIAL: NCT05080712
Title: Progression of Atrial Fibrillation in the Young
Acronym: PRAY
Status: Recruiting | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Principal Investigator, Piotr Sobocinski Doliwa, Principal Investigator, Karolinska Institutet
Other Study IDs: 2021-00992
Record Dates: First submitted 2021-09-23; First posted 2021-10-18 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; progression; left atrial function
MeSH Terms: conditions — Atrial Fibrillation; Disease Progression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to investigate the presence and magnitude of structural changes of the heart and their long-term development in young patients with atrial Fibrillation (AF), studied by echocardiographic measurements and plasma biomarkers and their association to AF burden, studied using long-term ECG

DETAILED DESCRIPTION:
100 patients with symptomatic Atrial Fibrillation diagnosis are included. Diagnosis is set either at the index visit or within 12 months before inclusion. . The follow up period is 5 years. Patients presenting with AF in connection with acute infection, acute cardiac ischemia, surgery or thyroid disease are excluded. Further, AF patients with cardiomyopathies, known genetic diseases and congenital cardiac abnormalities are also excluded.

At inclusion patients undergo an in-depth interview regarding comorbidities, medication, previous treatments related to the AF diagnosis. In addition, baseline data for weight and height are collected.

In connection to inclusion the patients are asked leave venous bloodwork (Na, K, Creatinine, plasma Glucose and NTproB-Type Natriuretic Peptide). An echocardiographic exam is performed according to a prespecified protocol with special emphasis on the left atrial function and anatomy. This is followed by a continuous ECG recording for 14 days using BioTel ePatch. The ECG patch is later returned to a core facility by mail.

The patients´ are followed for five years and are asked to leave bloodwork and perform a 14-day ECG recording yearly. After these exams, a follow up phone call is placed to the patient aimed at documenting clinical progress related to symptoms, treatment and interventions. After 5 years follow up patients undergo a follow up echocardiographic exam in addition to yearly bloodwork and ECG recording. The patients´ clinical symptoms are treated at the clinician´s discretion according to current guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Atrial fibrillation
* Diagnosis of atrial fibrillation within one year of inclusion

Exclusion Criteria:

* Duration of atrial fibrillation over one year.
* Acute stressor for atrial fibrillation such as: acute ischemic heart disease or infection

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with new onset atrial fibrillation within 12 months from inclusion
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-09-25 (Actual); Primary Completion 2027-12-20 (Estimated); Study Completion 2027-12-20 (Estimated)

PRIMARY OUTCOMES:
Development of atrial fibrillation burden | change from baseline at 5 years
  Change in burden of atrial fibrillation expressed as proportion of arrhythmia present on long-term ECG yearly

SECONDARY OUTCOMES:
Development of humoral measures of hemodynamic status | Change from baseline at 5 years
  Change in levels of plasma-N-terminal pro brain natriuretic peptide yearly (ng)
Development of atrial electrocardiographic status | Change from baseline at 5 years
  Change in number of supraventricular ectopic beats per 24 h on long-term ECG Yearly
Development of supraventricular ectopies | Change from baseline at 5 years
  Change in numbers of supraventricular tachycardia runs of at least 20 beats per 24 h on long-term ECG yearly
Development of atrial fibrillation incident | Change from baseline at 5 years
  Change in numbers of atrial fibrillation episodes per 24 h on long-term ECG yearly
Development of echocardiographic status | Change from baseline at 5 years
  Change in the left atrial volume indexed (ml/m2)
Development of left atrial systolic function by echocardiography | Change from baseline at 5 years
  Change in left atrial strain (%)
Development of left atrial volume by echocardiography | Change from baseline at 5 years
  Change in left ventricular volume indexed (ml/m2)
Development of left ventricular systolic function by echocardiographic | Change from baseline at 5 years
  Change in left ventricular ejection fraction (%)

CONTACTS AND LOCATIONS:
Overall Officials: Piotr Sobocinski Doliwa, MD, PhD, Study Chair — Karolinska Institutet Danderyds University Hospital
Locations (1):
- Danderyd Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided